CLINICAL TRIAL: NCT05475652
Title: The Influence of Manual Therapy Applied to the Cervical Spine (Versus Light Touch) in the Prevention of Balance Disorders in the Elderly: a Randomized Controlled Trial
Brief Title: The Influence of Manual Therapy Applied to the Cervical Spine in the Prevention of Balance Disorders in the Elderly
Acronym: ManEq
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EZUS-LYON 1 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 002B2019
Record Dates: First submitted 2022-05-20; First posted 2022-07-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Balance, Postural; Gait; Elderly
Keywords: senior;; gait; neck; myofascial release
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (ligth touch) (Sham Comparator): Placebo intervention composed of light touch treatment on the cervical spine.
  Interventions: Other: Placebo intervention
- Manual therapy (Experimental): Manual therapy applied to the cervical spine.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — The manual therapy intervention is performed twice on the experimental group, once on day 0 (D0) and the second time on day 7 (D7). This intervention consists of a manual therapy protocol (base on myofascial release) applied to the cervical spine. Protocol consists of succession of techniques: suboccipital decompression, disengagement of Cervical 0-1-2,vibratory stimulation at C4 level and myofascial release technique of the cervical aponeuroses. Outcomes are evaluated before and after intervention.The same schedule will be reproduced on D7. On D21, only one assessment will be done at the beginning of the session.
  Arms: Manual therapy
Other: Placebo intervention — The Sham group receives placebo treatment twice (D0 and D7). This placebo treatment also called "light touch" treatment consists of applying light pressure with broad support from both hands on either side of the joint, in contact with the skin, without equal bone pressure or therapeutic intention, for a duration comparable to that of manual therapy. Outcomes are evaluation before and after placebo intervention. The same schedule will be reproduced at D7. On D21, only one assessment will be done at the beginning of the session and a manual therapy treatment on the cervical spine is provided to balance access to care in the two group
  Arms: Sham (ligth touch)

SUMMARY:
Falling is a major trauma that can occur with aging, leading to very significant psychological and physical health effects with financial and societal consequences. It is therefore essential to explore therapeutic treatments that can reduce this risk. Some recognized effective treatments exist, concerning in particular the re-education of the muscles of the lower limbs. However, to our knowledge, none of them focus on the cervical spine although the latter is located at an essential physiological crossroads. Manual therapy, which has already demonstrated its impact on pain and balance parameters in the elderly, could be a painless and non-invasive tool of choice in addressing this problem.

DETAILED DESCRIPTION:
The main hypothesis of the present study is therefore that manual therapy applied to the cervical spine may have a beneficial impact on the balance and motor performance of seniors. The study also aims to propose an assessment of the physical parameters of balance, in order to validate the contribution of the cervical spine in compensatory mechanisms.

To do so, an interventional study was designed, monocentric, prospective, controlled, randomized double-blind (patient and evaluator performing the measurements). The experiment will take place over three measurement periods on D0, D7 and D21.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older, of either sex
* Autonomous, able to walk ten meters alone without walking aid
* Able to understand instructions necessary for the correct performance of the measurements.

Exclusion Criteria:

* Patients suffering from a locomotor handicap or severe chronic progressive pathologies preventing the protocol from being carried out correctly
* Patient who has an history of surgery - fracture - dislocation of the cervical spine
* Patient who has cognitive impairments (Mini Mental Statement <20)
* Patient who has life expectancy less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change of SPPB (Short Physical Performance Battery test) score at day 0 after 1 intervention | at Day 0 before and immediately after intervention in both groups
  The subject will then be asked to stand up and perform the different steps of the Short Physical Performance Battery test following the instructions of the evaluator, leading to a score between 0 (worse score) and 12 (best score)
change of SPPB (Short Physical Performance Battery test) score at day 7 after a second intervention | at Day 7 before and immediately after intervention in both groups
  The subject will then be asked to stand up and perform the different steps of the Short Physical Performance Battery test following the instructions of the evaluator, leading to a score between 0 (worse score) and 12 (best score)
SPPB (Short Physical Performance Battery test) score at day 21 | at Day 21 in both groups before the intervention for sham group
  The subject will then be asked to stand up and perform the different steps of the Short Physical Performance Battery test following the instructions of the evaluator, leading to a score between 0 (worse score) and 12 (best score)
change of walking speed at day 0 after 1 intervention | at Day 0 before and immediately after intervention in both groups
  The subject will performed a 4m gait measurement
change of walking speed at day 7 after a second intervention intervention | at Day 7 before and immediately after intervention in both groups
  The subject will performed a 4m gait measurement
walking speed at day 21 | at Day 21 in both groups, before the intervention for sham group
  The subject will performed a 4m gait measurement

SECONDARY OUTCOMES:
change in Heart Rate Variability at day 0 after 1 intervention | at Day 0 before and immediately after intervention in both groups
  Participants will be equipped with a heart rate monitor (Polar RS800) and a heart belt to collect HRV. The watch will be placed on the subjects' wrists and the belt on the chest (under the pectoral muscles for men and under the bra for women). The skin under the sensor will be slightly moistened to ensure good electrical contact and to avoid artifacts. The belt must be tight enough to ensure that the sensor is in perfect contact with the skin but must remain comfortable. Thus, a total recording time of 5 minutes, in the supine position and with spontaneous breathing, will be performed on each patient.
change in Heart Rate Variability at day 7 after the second intervention | at Day 7 before and immediately after intervention in both groups
  Participants will be equipped with a heart rate monitor (Polar RS800) and a heart belt to collect HRV. The watch will be placed on the subjects' wrists and the belt on the chest (under the pectoral muscles for men and under the bra for women). The skin under the sensor will be slightly moistened to ensure good electrical contact and to avoid artifacts. The belt must be tight enough to ensure that the sensor is in perfect contact with the skin but must remain comfortable. Thus, a total recording time of 5 minutes, in the supine position and with spontaneous breathing, will be performed on each patient.
Heart Rate Variability at day 21 | at Day 21 before the intervention for sham group
  Participants will be equipped with a heart rate monitor (Polar RS800) and a heart belt to collect HRV. The watch will be placed on the subjects' wrists and the belt on the chest (under the pectoral muscles for men and under the bra for women). The skin under the sensor will be slightly moistened to ensure good electrical contact and to avoid artifacts. The belt must be tight enough to ensure that the sensor is in perfect contact with the skin but must remain comfortable. Thus, a total recording time of 5 minutes, in the supine position and with spontaneous breathing, will be performed on each patient.
change in cervical range of motion at day 0 after 1 intervention | at Day 0 before and immediately after intervention in both groups
  the patients will be seated in a neutral position, with their backs against the back of the chair, and will perform the cervical range of motion tests. For this, the experimenter will use the anatomical points previously identified: ear tragus, chin symphysis, anterior angle of the acromion, sternal incisure. The subject will be asked to perform movements of flexion, extension, right rotation, left rotation, right tilt, and left tilt, returning to the neutral position each time. All movements will be performed 3 times. The measurement will retain the difference between the neutral position and the maximum position of the movement
change in cervical range of motion at day 7 after the second intervention | at Day 7 before and immediately after intervention in both groups
  the patients will be seated in a neutral position, with their backs against the back of the chair, and will perform the cervical range of motion tests. For this, the experimenter will use the anatomical points previously identified: ear tragus, chin symphysis, anterior angle of the acromion, sternal incisure. The subject will be asked to perform movements of flexion, extension, right rotation, left rotation, right tilt, and left tilt, returning to the neutral position each time. All movements will be performed 3 times. The measurement will retain the difference between the neutral position and the maximum position of the movement
cervical range of motion at day 21 | at Day 21 before the intervention for sham group
  the patients will be seated in a neutral position, with their backs against the back of the chair, and will perform the cervical range of motion tests. For this, the experimenter will use the anatomical points previously identified: ear tragus, chin symphysis, anterior angle of the acromion, sternal incisure. The subject will be asked to perform movements of flexion, extension, right rotation, left rotation, right tilt, and left tilt, returning to the neutral position each time. All movements will be performed 3 times. The measurement will retain the difference between the neutral position and the maximum position of the movement
change in cervical muscle strength at day 0 after 1 intervention | at Day 0 before and immediately after intervention in both groups
  the cervical strength tests will be performed seated too, using a manual dynamometer (Micro FET2, Hoggan, Salt Lake City, USA). To obtain the maximum isometric force of the neck muscles in the 6 movements, a "make test" will be performed: the experimenter will resist the subject's force without trying to exceed it. The subject will be asked to perform progressively and as hard as possible, from the neutral position, a flexion movement (resistance applied under the chin), an extension movement (resistance applied to the back of the occiput), a right and left rotation movement (resistance applied along the horizontal side of the right and left mandibles), and a right and left tilt movement (resistance applied above the right and left ears).
change in cervical muscle strength at day 7 after the second intervention | at Day 7 before and immediately after intervention in both groups
  the cervical strength tests will be performed seated too, using a manual dynamometer (Micro FET2, Hoggan, Salt Lake City, USA). To obtain the maximum isometric force of the neck muscles in the 6 movements, a "make test" will be performed: the experimenter will resist the subject's force without trying to exceed it. The subject will be asked to perform progressively and as hard as possible, from the neutral position, a flexion movement (resistance applied under the chin), an extension movement (resistance applied to the back of the occiput), a right and left rotation movement (resistance applied along the horizontal side of the right and left mandibles), and a right and left tilt movement (resistance applied above the right and left ears).
cervical muscle strength at day 21 | at Day 21 before the intervention for sham group
  the cervical strength tests will be performed seated too, using a manual dynamometer (Micro FET2, Hoggan, Salt Lake City, USA). To obtain the maximum isometric force of the neck muscles in the 6 movements, a "make test" will be performed: the experimenter will resist the subject's force without trying to exceed it. The subject will be asked to perform progressively and as hard as possible, from the neutral position, a flexion movement (resistance applied under the chin), an extension movement (resistance applied to the back of the occiput), a right and left rotation movement (resistance applied along the horizontal side of the right and left mandibles), and a right and left tilt movement (resistance applied above the right and left ears).
change in quadriceps strength at day 0 after 1 intervention | At Day 0 before and immediately after intervention in both groups
  to measure the maximal isometric extension force of the dominant quadriceps by applying the dynamometer to the lower tibia and requesting leg extension from a 90° flexion position
change in quadriceps strength at day 7 after the second intervention | At Day 7 before and immediately after intervention in both groups
  to measure the maximal isometric extension force of the dominant quadriceps by applying the dynamometer to the lower tibia and requesting leg extension from a 90° flexion position
quadriceps strength at day 21 | At Day 21 before the intervention for sham group
  to measure the maximal isometric extension force of the dominant quadriceps by applying the dynamometer to the lower tibia and requesting leg extension from a 90° flexion position
change in static posturography at day 0 after 1 intervention | At Day 0 before and immediately after intervention in both groups
  the static posturography test will be performed under standard conditions using the WIN-POSTURO platform (Medicapteur, Balma, France) allowing the measurement of displacements of the center of pressure in a static standing position at a frequency of 40 Hz for 25.6 seconds
  . The measurement will be repeated 3 times. The data collected will be processed using WIN-POSTURO software (Medicapteur, Balma, France)
change in static posturography at day 7 after the second intervention | At Day 7 before and immediately after intervention in both groups
  the static posturography test will be performed under standard conditions using the WIN-POSTURO platform (Medicapteur, Balma, France) allowing the measurement of displacements of the center of pressure in a static standing position at a frequency of 40 Hz for 25.6 seconds
  . The measurement will be repeated 3 times. The data collected will be processed using WIN-POSTURO software (Medicapteur, Balma, France)
static posturography at day 21 | At Day 21 before the intervention for sham group
  the static posturography test will be performed under standard conditions using the WIN-POSTURO platform (Medicapteur, Balma, France) allowing the measurement of displacements of the center of pressure in a static standing position at a frequency of 40 Hz for 25.6 seconds
  . The measurement will be repeated 3 times. The data collected will be processed using WIN-POSTURO software (Medicapteur, Balma, France)
change in plantar support at day 0 after 1 intervention | At Day 0 before and immediately after intervention in both groups
  The subject will perform the 4 m gait measurement part (which will measure walking speed) equipped with W-INSHOE plantar sensors (Medicapteur, Balam, France) which will be analyzed using the software of the same name. The sensors are attached to the skin with hypoallergenic tape
change in plantar support at day 7 after the second intervention | At Day 7 before and immediately after intervention in both groups
  The subject will perform the 4 m gait measurement part (which will measure walking speed) equipped with W-INSHOE plantar sensors (Medicapteur, Balam, France) which will be analyzed using the software of the same name. The sensors are attached to the skin with hypoallergenic tape
plantar support at day 21 | At Day 21 before the intervention for sham group
  The subject will perform the 4 m gait measurement part (which will measure walking speed) equipped with W-INSHOE plantar sensors (Medicapteur, Balam, France) which will be analyzed using the software of the same name. The sensors are attached to the skin with hypoallergenic tape

CONTACTS AND LOCATIONS:
Overall Officials: Laurianne PINLOCHE, MD, Principal Investigator — Laboratoire Interuniversitaire de Biologie de la Motricité
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinloche L, Souvignet S, Germain M, Monteil K, Hautier C. The short-term effect of a myofascial protocol versus light touch applied to the cervical spine towards the prevention of balance disorders in the elderly: protocol of a randomised controlled trial. Chiropr Man Therap. 2022 Aug 31;30(1):33. doi: 10.1186/s12998-022-00446-0. PMID 36045446